CLINICAL TRIAL: NCT01826149
Title: The Effect of Propofol on Tissue Doppler Imaging of Mitral Valve Annular Velocity During Remifentanil-based Cardiac Anesthesia
Brief Title: Propofol Effects on Mitral Valve Annular Velocity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor, Konkuk University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: KUH1160053
Record Dates: First submitted 2013-03-22; First posted 2013-04-08 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Valvular Heart Disease; Coronary Artery Disease
MeSH Terms: conditions — Heart Valve Diseases; Coronary Artery Disease | interventions — Propofol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Propofol 1.0mcg (Experimental): Propofol dosage titration, comparison of the effect of different concentration of propofol to the myocardial performances, namely at 1.0mcg/ml using target controlled infusion.
  Interventions: Drug: Propofol 1.0mcg
- Propofol 2.0mcg (Experimental): Propofol dosage titration, comparison of the effect of different concentration of propofol to the myocardial performances, namely at 2.0mcg/ml using target controlled infusion.
  Interventions: Drug: Propofol 2.0mcg
- Propofol 3.0mcg (Experimental): Propofol dosage titration, comparison of the effect of different concentration of propofol to the myocardial performances, namely at 3.0mcg/ml using target controlled infusion.
  Interventions: Drug: Propofol 3.0mcg

INTERVENTIONS:
Drug: Propofol 1.0mcg — Propofol dosage titration to achieve effect site concnetration at 1.0 mcg/ml using target controlled infusion.
  Other Names: Fresofol (2% propofol, Fresinius Kabi)
  Arms: Propofol 1.0mcg
Drug: Propofol 2.0mcg — Propofol dosage titration to achieve effect site concnetration at 2.0 mcg/ml using target controlled infusion.
  Other Names: Fresofol (2% propofol, Fresinius Kabi)
  Arms: Propofol 2.0mcg
Drug: Propofol 3.0mcg — Propofol dosage titration to achieve effect site concnetration at 3.0 mcg/ml using target controlled infusion
  Other Names: Fresofol (2% propofol, Fresinius Kabi)
  Arms: Propofol 3.0mcg

SUMMARY:
The purpose of this study is primarily to determine the effects of propofol at different concentration on the mitral valve annulus by using Tissue Doppler Imaging

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effects of different concentration of propofol on patients who are undergoing cardiac surgery. The patients will receive infusion remifentanil 0.5mcg/kg/min with different target-site propofol concentration namely 1.0ng/ml, 2.0ng/ml and 3.0ng/ml. Tissue Doppler Imaging by transesophageal echocardiography will be done to assess the changes in cardiac function.

ELIGIBILITY:
Inclusion Criteria:

patients undergoing cardiac surgery

Exclusion Criteria:

low ejection fraction < 50% on transthoracic echocardiography atrial fibrillation pacemaker pericardial and infiltrative myocardial disease mitral annular calcification, surgical rings, prosthetic mitral valve lateral left ventricular wall motion abnormality oesophageal abnormality history of extensive radiation to the mediastinum upper gastrointestinal bleeding

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change of systolic mitral valve annular velocity (S') | 10 min after achieving 3 different propofol concentrations
  To examine the effect of Propofol at different effect-site concentration ( 1.0 ng/ml, 2.0 ng/ml and 3.0 ng/ml) on S' (systolic mitral valve annular velocity) during remifentanil-based anesthesia.

SECONDARY OUTCOMES:
Early diastolic mitral valve annular velocity (e') | 10 min after achieving 3 different propofol concentrations
late diastolic (atrial contractile) mitral valve annular velocity (a') | 10 min after achieving 3 different propofol concentrations
ejection fraction | 10 min after achieving 3 different propofol concentrations
phenylephrine infusion rate | 10 min after achieving 3 different propofol concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Tae-yop Kim, MD, PhD, Principal Investigator — Konkuk University Medical Center, Seoul, Korea, Republic of
Locations (1):
- Konkuk University Medical Center, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Bang JY, Kim S, Choi BM, Kim TY. Pharmacodynamic Analysis of the Influence of Propofol on Left Ventricular Long-Axis Systolic Performance in Cardiac Surgical Patients. J Korean Med Sci. 2019 Apr 29;34(16):e132. doi: 10.3346/jkms.2019.34.e132. PMID 31020819